CLINICAL TRIAL: NCT02906670
Title: An Open-label, Multicenter, Phase 1a/2a Trial Investigating the Safety, Tolerability and Antitumor Activity of Multiple Doses of Sym013, a mAb Mixture Targeting EGFR, HER2 and HER3, in Patients With Advanced Epithelial Malignancies
Brief Title: Sym013 (Pan-HER) in Patients With Advanced Epithelial Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sym013-01
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Oncology
Keywords: Epithelial malignancies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- 1 mg/kg Q1W (Experimental): Phase 1a: Patients are administered a weekly dose of 1 mg/kg of Sym013 until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Interventions: Drug: Sym013
- 2 mg/kg Q1W (Experimental): Phase 1a: Patients are administered a weekly dose of 2 mg/kg of Sym013 until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Interventions: Drug: Sym013
- 4 mg/kg Q1W (Experimental): Phase 1a: Patients are administered a weekly dose of 4 mg/kg of Sym013 until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Interventions: Drug: Sym013
- 6 mg/kg Q1W + Prophylaxis (Experimental): Phase 1a: Patients are administered a weekly dose of 6 mg/kg of Sym013 + premedication until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Interventions: Drug: Sym013
- 9 mg/kg Q1W + Prophylaxis (Experimental): Phase 1a: Patients are administered a weekly dose of 9 mg/kg of Sym013 + premedication until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Interventions: Drug: Sym013
- 6 mg/kg Q2W (Experimental): Phase 1a: Patients are administered a dose of 6 mg/kg of Sym013 every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Interventions: Drug: Sym013
- 9 mg/kg Q2W (Experimental): Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Interventions: Drug: Sym013
- 9 mg/kg Q2W + Prophylaxis (Experimental): Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Interventions: Drug: Sym013
- 12 mg/kg Q2W + Prophylaxis (Experimental): Phase 1a: Patients are administered a dose of 12 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Interventions: Drug: Sym013
- 15 mg/kg Q2W + Prophylaxis (Experimental): Phase 1a: Patients are administered a dose of 15 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Interventions: Drug: Sym013
- Phase 2a Dose-Expansion Cohort A (Experimental): Part 2 is a Phase 2a dose-expansion with Sym013 at the RP2D and regimen. One (1) of 4 tumor types to be evaluated in this arm of the trial will be selected based upon findings from Part 1, additional preclinical data, and additional clinical data available at that time from other agents inhibiting these targets.
  Interventions: Drug: Sym013
- Phase 2a Dose-Expansion Cohort B (Experimental): Part 2 is a Phase 2a dose-expansion with Sym013 at the RP2D and regimen. One (1) of 4 tumor types to be evaluated in this arm of the trial will be selected based upon findings from Part 1, additional preclinical data, and additional clinical data available at that time from other agents inhibiting these targets.
  Interventions: Drug: Sym013
- Phase 2a Dose-Expansion Cohort C (Experimental): Part 2 is a Phase 2a dose-expansion with Sym013 at the RP2D and regimen. One (1) of 4 tumor types to be evaluated in this arm of the trial will be selected based upon findings from Part 1, additional preclinical data, and additional clinical data available at that time from other agents inhibiting these targets.
  Interventions: Drug: Sym013
- Phase 2a Dose-Expansion Cohort D (Experimental): Part 2 is a Phase 2a dose-expansion with Sym013 at the RP2D and regimen. One (1) of 4 tumor types to be evaluated in this arm of the trial will be selected based upon findings from Part 1, additional preclinical data, and additional clinical data available at that time from other agents inhibiting these targets.
  Interventions: Drug: Sym013

INTERVENTIONS:
Drug: Sym013 — Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
  Other Names: Pan-HER

SUMMARY:
This is the first study to test Sym013 (Pan-HER) in humans. The primary purpose of this study is to see if Sym013 is safe and effective for patients with advanced epithelial malignancies without available therapeutic options.

DETAILED DESCRIPTION:
This is an open-label, multicenter trial composed of 2 parts in which Sym013 will be evaluated when administered by intravenous infusion in patients with advanced epithelial malignancies without available therapeutic options.

Part 1 is a Phase 1a dose-escalation evaluating weekly (Q1W) and every second week (Q2W) schedules of administration in separate dose-escalation cohorts to determine the recommended phase 2 dose (RP2D) and regimen of Sym013.

Part 2 is a Phase 2a dose-expansion at the RP2D and regimen. Four (4) dose-expansion cohorts will be evaluated in this part of the trial and will be selected based upon findings from Part 1, additional preclinical data, and additional clinical data available at that time from other agents inhibiting these targets. Patients will be entered, depending upon either a defined molecular profile or profiles, or their underlying malignancy, to 1 of 4 corresponding expansion cohorts: Cohort A, Cohort B, Cohort C, or Cohort D.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria all patients, Part 1 and Part 2:

* Male or female, at least 18 years of age at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Life expectancy >3 months assessed during Screening
* Documented (histologically- or cytologically-proven) epithelial malignancy that is locally advanced or metastatic, having received all therapy known to confer clinical benefit

Additional inclusion criteria applicable to Part 2 ONLY:

* Epithelial malignancy (tumor types to be determined), measurable according to RECIST v1.1 that has been confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) within 4 weeks prior to C1/D1
* Willingness to undergo a pre-and post-dosing biopsy (total of 2 biopsies) from primary or metastatic tumor site(s) considered safe for biopsy

Exclusion Criteria:

* Any antineoplastic agent for the primary malignancy (standard or investigational) without delayed toxicity within 4 weeks or 5 plasma half-lives (whichever is shortest) prior to C1/D1, except nitrosoureas and mitomycin C within 6 weeks prior to C1/D1.
* Part 2 ONLY: Radiotherapy against target lesions within 4 weeks prior to C1/D1, unless there is documented progression of the lesion following radiotherapy
* Immunosuppressive or systemic hormonal therapy (>10 mg daily prednisone equivalent) within 2 weeks prior to C1/D1 with exceptions
* Use of hematopoietic growth factors within 2 weeks prior to C1/D1
* Active second malignancy or history of another malignancy within the last 3 years, with allowed exceptions
* Central nervous system (CNS) malignancies including:

  1. Primary malignancies of the CNS
  2. Known, untreated CNS or leptomeningeal metastases, or spinal cord compression; patients with any of these not controlled by prior surgery or radiotherapy, or symptoms suggesting CNS metastatic involvement for which treatment is required
* Inadequate recovery from an acute toxicity associated with any prior antineoplastic therapy
* Major surgical procedure within 4 weeks prior to C1/D1 or inadequate recovery from any prior surgical procedure
* Non-healing wounds on any part of the body
* Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks prior to C1/D1, unless adequately treated and stable
* Active uncontrolled bleeding or a known bleeding diathesis
* Significant gastrointestinal abnormalities
* Significant cardiovascular disease or condition
* Abnormal hematologic, renal or hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berlin J, Tolcher AW, Ding C, Whisenant JG, Horak ID, Wood DL, Nadler PI, Hansen UH, Lantto J, Skartved NJO, Pedersen MW, Patnaik A. First-in-human trial exploring safety, antitumor activity, and pharmacokinetics of Sym013, a recombinant pan-HER antibody mixture, in advanced epithelial malignancies. Invest New Drugs. 2022 Jun;40(3):586-595. doi: 10.1007/s10637-022-01217-7. Epub 2022 Feb 3. PMID 35113285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were only recruited for Part 1; a recommended Phase 2 dose (RP2D) could not be established and the part 2 cohorts A, B, C and were not initiated.
Groups:
- 1 mg/kg Q1W: Phase 1a: Patients are administered a weekly dose of 1 mg/kg of Sym013 for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
- 2 mg/kg Q1W: Phase 1a: Patients are administered a weekly dose of 2 mg/kg of Sym013 for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
- 4 mg/kg Q1W: Phase 1a: Patients are administered a weekly dose of 4 mg/kg of Sym013 for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
- 6 mg/kg Q1W + Prophylaxis: Phase 1a: Patients are administered a weekly dose of 6 mg/kg of Sym013 + premedication for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 9 mg/kg Q1W + Prophylaxis: Phase 1a: Patients are administered a weekly dose of 9 mg/kg of Sym013 + premedication for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 6 mg/kg Q2W: Phase 1a: Patients are administered 6 mg/kg of Sym013 every second week for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
- 9 mg/kg Q2W: Phase 1a: Patients are administered 9 mg/kg of Sym013 every second week for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
- 9 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered 9 mg/kg of Sym013 every second week for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 12 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered 12 mg/kg of Sym013 every second week for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 15 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered 15 mg/kg of Sym013 every second week for 4 weeks until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
Period: Cohort 1, QW
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Radiological Progression | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2, QW
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Radiological Progression | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3, QW
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Radiological Progression | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Clinical Benefit | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4, Q2W
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Radiological Progression | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Cohort 5, Q2W
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
Not completed — Radiological Progression | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Clinical Benefit | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Cohort 5P, Q2W
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Radiological Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Cohort 6P, Q2W
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Radiological Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Period: Cohort 4P, QW
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Radiological Progression | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 7P, Q2W
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — More than 3 Dose-reduction of Pan-Her | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Cohort 5P, QW
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Started | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Radiological Progression | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 mg/kg Q1W: Phase 1a: Patients are administered a weekly dose of 1 mg/kg of Sym013 until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
- 2 mg/kg Q1W: Phase 1a: Patients are administered a weekly dose of 2 mg/kg of Sym013 until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
- 4 mg/kg Q1W: Phase 1a: Patients are administered a weekly dose of 4 mg/kg of Sym013 until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
- 6 mg/kg Q1W + Prophylaxis: Phase 1a: Patients are administered a weekly dose of 6 mg/kg of Sym013 + premedication until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 9 mg/kg Q1W + Prophylaxis: Phase 1a: Patients are administered a weekly dose of 9 mg/kg of Sym013 + premedication until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 6 mg/kg Q2W: Phase 1a: Patients are administered a dose of 6 mg/kg of Sym013 every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
- 9 mg/kg Q2W: Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
- 9 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 12 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 12 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- 15 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 15 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
- Total: Total of all reporting groups
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Total
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 7 | 3 | 4 | 3 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 2 | 1 | 2 | 6 | 1 | 1 | 2 | 20
  >=65 years | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 | 57.0 | 59.3 (9.74) | 58.0 (6.08) | 63.3 (11.24) | 56.0 (12.12) | 51.6 (11.59) | 67.3 (10.02) | 63.8 (13.77) | 59.7 (8.02) | 58.7 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 3 | 1 | 1 | 12
  Male | 1 | 1 | 3 | 3 | 1 | 2 | 4 | 0 | 3 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 6
  Not Hispanic or Latino | 1 | 1 | 3 | 1 | 3 | 3 | 6 | 2 | 4 | 2 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
  White | 1 | 1 | 3 | 3 | 2 | 2 | 6 | 2 | 4 | 3 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 4 | 3 | 3 | 3 | 7 | 3 | 4 | 3 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 36.2 | 26.30 | 27.45 (7.543) | 26.00 (2.893) | 26.93 (2.409) | 27.13 (2.122) | 26.84 (5.828) | 24.03 (6.584) | 21.98 (1.981) | 31.83 (9.178) | 26.75 (5.575)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Assess the Safety and Tolerability of Sym013 When Administered Either Q1W or Q2W to Separate Dose-escalation Cohorts of Patients.
Description: Assess the occurrence of dose-limiting toxicities (DLTs) during Cycle 1 of Sym013 administration.
Time Frame: 24 months
Population: Pts 84001-007 (9mg/kg Q2W) and 84002-01 (12 mg/kg +P Q2W) did not complete C1 and hence is not considered eligible for DLT assessments.
Measure: Count of Participants; unit: Participants
Groups:
- 12 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 12 mg/kg of Sym013 + premedication every second until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 6 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2

2. Primary Outcome: Part 2: Evaluate the Antitumor Effect of Sym013 When Administered at the RP2D and Regimen to Patients.
Description: No data were collected for this Outcome Measures as Part 2 of the trial was never initiated.
Time Frame: 24 months
Population: The outcome measure was not analyzed, because the study was stopped during Part 1 of the study before initiating Part 2 of the study for business reasons. No data were collected in Part 2
Arm/Group | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Part 1: Determine the RP2D and Regimen of Sym013.
Description: No RP2D or regimen of Sym013 was determined as the trial was prematurely terminated
Time Frame: 24 months
Population: No data were collected for this Outcome Measure for Parts 1 and 2
Groups:
- 6 mg/kg Q1W + Prophylaxis: Phase 1a: Patients are administered a weekly dose of 6 mg/kg of Sym013 + premedication until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Sym013: Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
- 9 mg/kg Q1W + Prophylaxis: Phase 1a: Patients are administered a weekly dose of 9 mg/kg of Sym013 + premedication until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Sym013: Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
- 9 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Sym013: Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
- 12 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 12 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Sym013: Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
- 15 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 15 mg/kg of Sym013 + premedication every second week until unacceptable toxicity, progressive disease, termination of the trial or patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Sym013: Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Parts 1 and 2: Evaluate the Immunogenicity of Sym013.
Description: Serum sampling to assess the potential for anti-drug antibody (ADA) formation was not analyzed as the trial was prematurely terminated
Time Frame: 42 months
Population: No data were collected for this Outcome Measure for Parts 1 and 2
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Parts 1 and 2: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC).
Description: Will be estimated using non-compartmental methods and actual time points.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours if Q2W
Population: No patients in the 15 mg/kg Q2W + Prophylaxis group proceeded to the 3rd dose Not all patients completed both PK profiles; thus lower patient number in 2nd PK profile than in 1st profile
Measure: Mean (Standard Deviation); unit: h*µg/mL
Groups:
- 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 (+ premedication) every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
  Sym013: Sym013 is a recombinant antibody mixture containing 6 humanized immunoglobulin G1 (IgG1) monoclonal antibodies (mAbs), which bind specifically to non-overlapping epitopes or domains on the epidermal growth factor receptor (EGFR), and the human epidermal growth factor receptors (HER) HER2 and HER3.
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 10 | 4 | 3 | 0 | 0 | 0 | 0
h*µg/mL
  Hu1277, 1st dose (1st PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | 22 | 270 (43) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 550 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | 280 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | 440 (24) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 8600 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |
  Hu1565, 1st dose (1st PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 1480 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | 2200 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 2900 (1100) | 3900 (670) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) |  |  |  |
  Hu4384, 1st dose (1st PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 750 (110) | 1200 (230) | 2100 (640) | 1000 (310) | 2200 (960) | 2600 (570) | 19000 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |
  Hu4517, 1st dose (1st PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 267 | 880 (130) | 1400 (320) | 2300 (680) | 1200 (250) | 2200 (690) | 2600 (710) | 17000 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |
  Hu5038, 1st dose (1st PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 860 (85) | 1200 (280) | 2000 (680) | 1100 (310) | 2000 (580) | 2500 (1000) | 13500 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |
  Hu5082, 1st dose (1st PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 628 | 2900 (230) | 3900 (1100) | 3900 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | 4000 (1500) | 6000 (1800) | 8900 (3700) | 19800 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |
  Hu1277, 3rd/4th dose (2nd PK profile), AUC: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1277, 3rd/4th dose (2nd PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 760 (300) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) |  |  |  |  |
  Hu1565, 3rd/4th dose (2nd PK profile), AUC: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1565, 3rd/4th dose (2nd PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 1300 (720) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 2100 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) |  |  |  |  |
  Hu4384, 3rd/4th dose (2nd PK profile), AUC: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4384, 3rd/4th dose (2nd PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 1600 (1000) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 1800 (570) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) |  |  |  |  |
  Hu4517, 3rd/4th dose (2nd PK profile), AUC: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4517, 3rd/4th dose (2nd PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | 340 | 1800 (1200) | 2100 (200) | 5600 (4600) | 1700 (400) | 2500 (1200) | 3100 (870) |  |  |  |  |
  Hu5038, 3rd/4th dose (2nd PK profile), AUC: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5038, 3rd/4th dose (2nd PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 1600 (870) | 1500 (470) | 4000 (3100) | 1800 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | 2500 (1200) | 4800 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |  |
  Hu5082, 3rd/4th dose (2nd PK profile), AUC: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5082, 3rd/4th dose (2nd PK profile), AUC | NA — Patient analyzed; not reportable due to not meeting the criteria for reporting (no apparent profile; to few data points) | 880 | 2600 (740) | 6800 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high) | 3800 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD | 9900 (2600) | 9700 (NA) — All patients analyzed; 1 patient fulfilled criteria for reporting; rest was not reportable due to not meeting the criteria for reporting (extrapolation per cent for AUC was to high), thus no SD |  |  |  |  |

6. Secondary Outcome: Parts 1 and 2: Maximum Concentration (Cmax) and Trough Concentration (Ctrough) - Mean Values.
Description: Will be derived from observed data.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours if Q2W
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis: Phase 1a: Patients are administered a dose of 9 mg/kg of Sym013 (+ premedication) every second week until unacceptable toxicity, progressive disease, termination of the trial or the patient decision to withdraw.
  Premedications for infusion-related reactions included glucocorticoids and an antihistamine (H1 antagonist) prior to each dose of Pan-HER from the beginning of the study. As of Protocol Amendment 5, additional premedications were added which included montelukast, dexamethasone, antihistamine (H2 antagonist), and acetaminophen.
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 10 | 4 | 3
µg/mL
  Hu1277, 1st dose (1st PK profile), Cmax | 0.78 | 1.8 | 10 (3.0) | 15 (3.1) | 23 (2.6) | 12 (2.5) | 20 (9.0) | 25 (3.7) | 66 (21)
  Hu1277, 1st dose (1st PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | 16 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit
  Hu1565, 1st dose (1st PK profile), Cmax | 3.2 | 4.9 | 21 (4.3) | 31 (5.6) | 44 (3.1) | 25 (3.9) | 43 (17) | 48 (6.3) | 130 (34)
  Hu1565, 1st dose (1st PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | 0.82 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit | 0.85 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | 50 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit
  Hu4384, 1st dose (1st PK profile), Cmax | 2.5 | 4.1 | 16 (6.2) | 22 (3.2) | 30 (2.3) | 16 (3.0) | 30 (11) | 31 (3.7) | 92 (45)
  Hu4384, 1st dose (1st PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | 0.32 | 0.59 (0.36) | 1.5 (0.9) | 3.3 (1.9) | NA (NA) — All patients analyzed; not reportable due to values below detection limit | 0.69 (0.55) | 1.4 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit | 19 (23)
  Hu4517, 1st dose (1st PK profile), Cmax | 3.0 | 4.7 | 17 (2.2) | 27 (4.5) | 36 (4.2) | 20 (2.9) | 37 (16) | 38 (3.9) | 110 (55)
  Hu4517, 1st dose (1st PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | 0.38 | 0.72 (0.31) | 1.4 (0.9) | 3.0 (1.5) | 0.43 (0.05) | 0.66 (0.22) | 0.61 (0.21) | 16 (22)
  Hu5038, 1st dose (1st PK profile), Cmax | 2.9 | 5.6 | 16 (2.3) | 24 (4.0) | 31 (2.4) | 18 (2.9) | 29 (12) | 34 (3.9) | 87 (32)
  Hu5038, 1st dose (1st PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | 0.79 (0.24) | 1.3 (1.1) | 2.8 (1.8) | NA (NA) — All patients analyzed; not reportable due to values below detection limit | 0.57 (0.24) | 0.86 (0.29) | 15 (19)
  Hu5082, 1st dose (1st PK profile), Cmax | 7.2 | 9.8 | 42 (6.5) | 55 (11) | 67 (6.3) | 39 (12) | 77 (32) | 89 (14) | 160 (45)
  Hu5082, 1st dose (1st PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | 0.92 | 4.8 (0.7) | 9.3 (6.3) | 16 (11) | 2.5 (2.2) | 4.3 (2.0) | 7.8 (3.7) | 34 (43)
  Hu1277, 3rd/4th dose (2nd PK profile), Cmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu1277, 3rd/4th dose (2nd PK profile), Cmax | 2.5 | 3.0 | 11 (1.3) | 17 (2.3) | 30 (6.6) | 13 (1.6) | 28 (11) | 29 (3.9) |
  Hu1277, 3rd/4th dose (2nd PK profile), Ctrough: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu1277, 3rd/4th dose (2nd PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit |
  Hu1565, 3rd/4th dose (2nd PK profile), Cmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu1565, 3rd/4th dose (2nd PK profile), Cmax | 9.5 | 7.0 | 22 (3.0) | 35 (8.7) | 54 (10) | 29 (5.7) | 57 (21) | 60 (8.8) |
  Hu1565, 3rd/4th dose (2nd PK profile), Ctrough: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu1565, 3rd/4th dose (2nd PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | 0.49 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit | 8.9 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit | 2.5 (0.3) | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit | NA (NA) — All patients analyzed; not reportable due to values below detection limit |
  Hu4384, 3rd/4th dose (2nd PK profile), Cmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu4384, 3rd/4th dose (2nd PK profile), Cmax | 8.3 | 6.1 | 17 (2.6) | 30 (4.2) | 48 (21) | 19 (3.6) | 37 (13) | 34 (3.6) |
  Hu4384, 3rd/4th dose (2nd PK profile), Ctrough: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu4384, 3rd/4th dose (2nd PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | 1.9 (0.8) | 6.6 (4.7) | 10 (7.0) | NA (NA) — All patients analyzed; not reportable due to values below detection limit | 1.5 (1.8) | NA (NA) — All patients analyzed; not reportable due to values below detection limit |
  Hu4517, 3rd/4th dose (2nd PK profile), Cmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu4517, 3rd/4th dose (2nd PK profile), Cmax | 8.4 | 7.5 | 19 (2.5) | 31 (8.1) | 57 (19) | 21 (0.8) | 43 (13) | 45 (5.6) |
  Hu4517, 3rd/4th dose (2nd PK profile), Ctrough: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu4517, 3rd/4th dose (2nd PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | 0.59 | 2.1 (0.9) | 4.9 (3.4) | 5.4 (1.0) | 0.66 (0.22) | 1.3 (1.1) | 0.75 (0.41) |
  Hu5038, 3rd/4th dose (2nd PK profile), Cmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu5038, 3rd/4th dose (2nd PK profile), Cmax | 7.7 | 8.3 | 18 (2.1) | 29 (4.0) | 44 (9.1) | 21 (4.1) | 42 (14) | 41 (3.9) |
  Hu5038, 3rd/4th dose (2nd PK profile), Ctrough: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu5038, 3rd/4th dose (2nd PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | NA — Patient analyzed; not reportable due to values below detection limit | 1.9 (0.4) | 3.8 (2.7) | 4.5 (1.9) | 0.81 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit | 1.4 (1.2) | 2.6 (NA) — All patients analyzed; only 1 result above level of detection, rest not reportable due to values below detection limit |
  Hu5082, 3rd/4th dose (2nd PK profile), Cmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu5082, 3rd/4th dose (2nd PK profile), Cmax | 10 | 15 | 47 (9.6) | 97 (42) | 82 (23) | 51 (6.8) | 99 (31) | 120 (21) |
  Hu5082, 3rd/4th dose (2nd PK profile), Ctrough: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0
  Hu5082, 3rd/4th dose (2nd PK profile), Ctrough | NA — Patient analyzed; not reportable due to values below detection limit | 1.9 | 7.1 (6.1) | 28 (16) | 31 (20) | 6.8 (6.8) | 6.2 (6.2) | 22 (22) |

7. Secondary Outcome: Parts 1 and 2: Time to Reach Maximum Concentration (Tmax).
Description: Will be derived from observed data. End of infusion was defined as time zero (0)
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours if Q2W
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 10 | 4 | 3 | 0 | 0 | 0 | 0
h
  Hu1277, 1st dose (1st PK profile), Tmax | 0 | 0 | 2.5 (1.9) | 2.0 (2.0) | 1.1 (1.0) | 0.69 (1.2) | 1.7 (1.9) | 0.91 (1.1) | 0.94 (1.6) |  |  |  |
  Hu1565, 1st dose (1st PK profile), Tmax | 0 | 0 | 2.5 (1.9) | 0.65 (1.1) | 2.3 (1.1) | 0.69 (1.2) | 1.9 (1.8) | 1.4 (1.0) | 2.2 (1.9) |  |  |  |
  Hu4384, 1st dose (1st PK profile), Tmax | 0 | 0 | 2.5 (1.9) | 0.65 (1.1) | 2.3 (1.1) | 0 (0) | 3.1 (5.4) | 1.3 (0.89) | 1.2 (2.1) |  |  |  |
  Hu4517, 1st dose (1st PK profile), Tmax | 0 | 0 | 2.5 (1.9) | 2.0 (2.0) | 1.1 (0.97) | 0 (0) | 1.3 (1.1) | 1.0 (1.1) | 0 (0) |  |  |  |
  Hu5038, 1st dose (1st PK profile), Tmax | 2.0 | 0 | 2.5 (1.9) | 2.0 (2.0) | 1.1 (0.97) | 0 (0) | 1.4 (1.3) | 1.0 (1.2) | 1.2 (2.1) |  |  |  |
  Hu5082, 1st dose (1st PK profile), Tmax | 0 | 0 | 2.5 (1.9) | 0.65 (1.1) | 1.1 (0.97) | 0.97 (1.2) | 1.1 (1.2) | 0.52 (1.0) | 6.4 (11) |  |  |  |
  Hu1277, 3rd/4th dose (2nd PK profile), Tmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1277, 3rd/4th dose (2nd PK profile), Tmax | 7.0 | 0 | 0.48 (0.96) | 0 (0) | 1.3 (2.3) | 0.97 (1.4) | 0.94 (1.0) | 0 (0) |  |  |  |  |
  Hu1565, 3rd/4th dose (2nd PK profile), Tmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1565, 3rd/4th dose (2nd PK profile), Tmax | 7.0 | 0 | 0 (0) | 0 (0) | 2.5 (2.2) | 0.67 (1.4) | 1.5 (2.0) | 1.7 (2.4) |  |  |  |  |
  Hu4384, 3rd/4th dose (2nd PK profile), Tmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4384, 3rd/4th dose (2nd PK profile), Tmax | 7.0 | 0 | 1.0 (2.0) | 0 (0) | 2.5 (2.2) | 0.97 (1.4) | 1.2 (2.1) | 0 (0) |  |  |  |  |
  Hu4517, 3rd/4th dose (2nd PK profile), Tmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4517, 3rd/4th dose (2nd PK profile), Tmax | 7.0 | 0 | 1.4 (1.8) | 1.3 (2.3) | 1.3 (2.3) | 0.97 (1.4) | 0.91 (1.5) | 0 (0) |  |  |  |  |
  Hu5038, 3rd/4th dose (2nd PK profile), Tmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5038, 3rd/4th dose (2nd PK profile), Tmax | 7.0 | 0 | 0.48 (0.96) | 0 (0) | 1.3 (2.3) | 0.97 (1.4) | 0.94 (1.0) | 0 (0) |  |  |  |  |
  Hu5082, 3rd/4th dose (2nd PK profile), Tmax: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5082, 3rd/4th dose (2nd PK profile), Tmax | 0 | 0 | 2.9 (2.4) | 1.9 (2.0) | 2.5 (2.2) | 0.97 (1.4) | 4.0 (8.3) | 0.95 (1.3) |  |  |  |  |

8. Secondary Outcome: Parts 1 and 2: Elimination Half-life (T½).
Description: Will be estimated using non-compartmental methods and actual time points
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours if Q2W
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: H
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 10 | 4 | 3 | 0 | 0 | 0 | 0
H
  Hu1277, 1st dose (1st PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 8.3 | 18 (4.1) | 26 (6.0) | 25 (5.8) | 21 (9.2) | 30 (20) | 39 (7.2) | 56 (18) |  |  |  |
  Hu1565, 1st dose (1st PK profile), T½ | 20 | 29 | 36 (5.8) | 29 (2.4) | 33 (10) | 35 (5.0) | 45 (14) | 52 (8.2) | 66 (24) |  |  |  |
  Hu4384, 1st dose (1st PK profile), T½ | 31 | 50 | 39 (5.6) | 51 (7.9) | 62 (12) | 47 (16) | 56 (19) | 73 (13) | 92 (48) |  |  |  |
  Hu4517, 1st dose (1st PK profile), T½ | 29 | 50 | 39 (4.7) | 43 (5.0) | 56 (9.8) | 59 (18) | 54 (15) | 55 (11) | 73 (32) |  |  |  |
  Hu5038, 1st dose (1st PK profile), T½ | 27 | 39 | 42 (4.0) | 42 (6.5) | 55 (11) | 50 (16) | 51 (12) | 54 (23) | 78 (44) |  |  |  |
  Hu5082, 1st dose (1st PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 53 | 66 (7.0) | 83 (30) | 96 (33) | 90 (33) | 96 (29) | 97 (34) | 93 (62) |  |  |  |
  Hu1277, 3rd/4th dose (2nd PK profile), T½: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1277, 3rd/4th dose (2nd PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 28 (9.6) | 37 (1.5) | 35 (7.7) | 27 (5.5) | 26 (7) | 31 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85); thus no SD |  |  |  |  |
  Hu1565, 3rd/4th dose (2nd PK profile), T½: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1565, 3rd/4th dose (2nd PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 20 | 43 (26) | 50 (22) | 43 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85); thus no SD | 39 (3.6) | 39 (8.3) | 48 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85); thus no SD |  |  |  |  |
  Hu4384, 3rd/4th dose (2nd PK profile), T½: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4384, 3rd/4th dose (2nd PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 25 | 69 (50) | 94 (25) | 152 (105) | 44 (3.7) | 84 (49) | 48 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85); thus no SD |  |  |  |  |
  Hu4517, 3rd/4th dose (2nd PK profile), T½: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4517, 3rd/4th dose (2nd PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 34 | 77 (50) | 64 (21) | 85 (27) | 70 (3.0) | 79 (35) | 61 (7.4) |  |  |  |  |
  Hu5038, 3rd/4th dose (2nd PK profile), T½: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5038, 3rd/4th dose (2nd PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 20 | 69 (40) | 62 (11) | 77 (28) | 59 (22) | 78 (41) | 64 (35) |  |  |  |  |
  Hu5082, 3rd/4th dose (2nd PK profile), T½: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5082, 3rd/4th dose (2nd PK profile), T½ | NA — Patient analyzed, not reportable due to not meeting the criteria for reporting (to few data points available, time span for lambda Z to short or R2 < 0.85) | 42 | 111 (90) | 137 (73) | 175 (71) | 119 (54) | 103 (30) | 177 (122) |  |  |  |  |

9. Secondary Outcome: Parts 1 and 2: Clearance (CL).
Description: Will be estimated using non-compartmental methods and actual time points.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours if Q2W
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W and 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis | Phase 2a Dose-Expansion Cohort A | Phase 2a Dose-Expansion Cohort B | Phase 2a Dose-Expansion Cohort C | Phase 2a Dose-Expansion Cohort D
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 10 | 4 | 3 | 0 | 0 | 0 | 0
mL/h/kg
  Hu1277, 1st dose (1st PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 9.8 | 1.6 (0.26) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 1.8 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | 2.3 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | 2.2 (0.12) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.19 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |
  Hu1565, 1st dose (1st PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.82 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | 0.82 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.72 (0.31) | 0.64 (0.11) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) |  |  |  |
  Hu4384, 1st dose (1st PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.63 (0.092) | 0.6 (0.12) | 0.53 (0.19) | 0.72 (0.19) | 0.59 (0.31) | 0.55 (0.12) | 0.093 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |
  Hu4517, 1st dose (1st PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.67 (0.11) | 0.64 (0.15) | 0.62 (0.22) | 0.77 (0.15) | 0.67 (0.29) | 0.69 (0.15) | 0.13 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |
  Hu5038, 1st dose (1st PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.60 (0.059) | 0.68 (0.17) | 0.62 (0.26) | 0.74 (0.18) | 0.64 (0.21) | 0.68 (0.24) | 0.14 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |
  Hu5082, 1st dose (1st PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.97 | 0.42 (0.033) | 0.49 (0.14) | 0.70 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | 0.50 (0.17) | 0.49 (0.13) | 0.46 (0.17) | 0.23 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |
  6Hu1277, 3rd/4th dose (2nd PK profile), CL: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  6Hu1277, 3rd/4th dose (2nd PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 1.4 (0.54) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) |  |  |  |  |
  Hu1565, 3rd/4th dose (2nd PK profile), CL: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu1565, 3rd/4th dose (2nd PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.79 (0.37) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.86 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) |  |  |  |  |
  Hu4384, 3rd/4th dose (2nd PK profile), CL: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4384, 3rd/4th dose (2nd PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.36 (0.16) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.63 (0.20) | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) |  |  |  |  |
  Hu4517, 3rd/4th dose (2nd PK profile), CL: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu4517, 3rd/4th dose (2nd PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.86 | 0.41 (0.20) | 0.42 (0.041) | 0.35 (0.29) | 0.54 (0.13) | 0.62 (0.29) | 0.59 (0.17) |  |  |  |  |
  Hu5038, 3rd/4th dose (2nd PK profile), CL: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5038, 3rd/4th dose (2nd PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.37 (0.15) | 0.55 (0.18) | 0.41 (0.31) | 0.42 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | 0.55 (0.25) | 0.32 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |  |
  Hu5082, 3rd/4th dose (2nd PK profile), CL: number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0
  Hu5082, 3rd/4th dose (2nd PK profile), CL | NA — Patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.69 | 0.49 (0.14) | 0.27 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | NA (NA) — All patients analyzed; not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high) | 0.48 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD | 0.29 (0.08) | 0.38 (NA) — All patients analyzed; only 1 patient fulfilled criteria for reporting, rest not reportable due to not meeting the criteria for reporting (parameter derived from AUC and extrapolation per cent for AUC was to high); thus no SD |  |  |  |  |

ADVERSE EVENTS:
Time Frame: All AEs will be recorded from signing of informed consent for participation in the trial. The recording period ends at the time of the 1 month follow-up Visit.
Arm/Group | 1 mg/kg Q1W | 2 mg/kg Q1W | 4 mg/kg Q1W | 6 mg/kg Q1W + Prophylaxis | 9 mg/kg Q1W + Prophylaxis | 6 mg/kg Q2W | 9 mg/kg Q2W | 9 mg/kg Q2W + Prophylaxis | 12 mg/kg Q2W + Prophylaxis | 15 mg/kg Q2W + Prophylaxis
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 0/3 | 0/3 | 1/3 | 0/7 | 0/3 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 0/3 | 1/3 | 1/3 | 3/7 | 1/3 | 2/4 | 2/7
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/4 | 3/3 | 3/3 | 3/3 | 7/7 | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg Q1W (N=1) | 2 mg/kg Q1W (N=1) | 4 mg/kg Q1W (N=4) | 6 mg/kg Q1W + Prophylaxis (N=3) | 9 mg/kg Q1W + Prophylaxis (N=3) | 6 mg/kg Q2W (N=3) | 9 mg/kg Q2W (N=7) | 9 mg/kg Q2W + Prophylaxis (N=3) | 12 mg/kg Q2W + Prophylaxis (N=4) | 15 mg/kg Q2W + Prophylaxis (N=7)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg Q1W (N=1) | 2 mg/kg Q1W (N=1) | 4 mg/kg Q1W (N=4) | 6 mg/kg Q1W + Prophylaxis (N=3) | 9 mg/kg Q1W + Prophylaxis (N=3) | 6 mg/kg Q2W (N=3) | 9 mg/kg Q2W (N=7) | 9 mg/kg Q2W + Prophylaxis (N=3) | 12 mg/kg Q2W + Prophylaxis (N=4) | 15 mg/kg Q2W + Prophylaxis (N=3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (10) | 2 (2) | 2 (9) | 2 (4) | 6 (9) | 1 (2) | 3 (5) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagai (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 3 (4) | 3 (7) | 2 (6) | 5 (8) | 1 (1) | 1 (1) | 2 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 3 (5) | 1 (3) | 3 (3) | 2 (4)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT02906670/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT02906670/SAP_001.pdf